CLINICAL TRIAL: NCT04556747
Title: Functional Outcome Response to Engaging Virtual Reality in Pediatric Patients (FOREVR Peds Study)
Brief Title: FOREVR Peds VR Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-2892
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Pain, Postoperative; Pain; Anxiety
MeSH Terms: conditions — Pain, Postoperative; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR - Distraction (Other)
  Interventions: Other: VR - Distraction
- VR - Biofeedback (Other)
  Interventions: Other: VR - Biofeedback

INTERVENTIONS:
Other: VR - Distraction — Participants will be instructed to use any application.
  Arms: VR - Distraction
Other: VR - Biofeedback — Participants will be instructed to use the Mindful Aurora application.
  Arms: VR - Biofeedback

SUMMARY:
To determine the feasibility and acceptability of using immersive virtual reality technologies to impact clinical outcomes (e.g., pain and anxiety) and medication utilization (e.g., narcotics) in pediatric patients with acute and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7to 21 years
* Able to read, understand, and speak English
* Patients in the immediate postoperative period with significant pain being followed by the Acute Pain Service (acute postoperative pain cohort); patients presenting in Same Day Surgery for peripheral IV placement or patients in the CBDI clinic presenting for peripheral IV placement or Port accessing (vascular access cohort); or patients admitted to CCHMC on the Medical Pain Service (chronic pain cohort), or sickle cell patients not on the MPS list.
* Patients who have undergone bone marrow transplantation or receiving chemotherapy experiencing pain from mucositis

Exclusion Criteria:

* Outside the age range (< 7 or > 21 years)
* History of developmental delays, uncontrolled psychiatric conditions, or neurological conditions (especially epilepsy and/or significant motion sickness/nausea/vomiting)
* History of vertigo, dizziness, and/or seizure disorder
* Conditions that would preclude the application of the VR glasses, such as surgeries of the head and neck

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Effect of VR-distraction on anxiety | Before 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-Distraction on anxiety | Immediately after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-Distraction on anxiety | 15 minutes after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-Distraction on anxiety | 30 minutes after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-Distraction on pain | Before 10 minute VR session.
  Pain scores will be collected. Pain will be rated using a numerical rating scale. Pain will be rated from 0 - 10. 0 meaning no pain 10 being severe pain
Effect of VR-Distraction on pain | Immediately after 10 minute VR session.
  Pain scores will be collected. Pain will be rated using a numerical rating scale. Pain will be rated from 0 - 10. 0 meaning no pain 10 being severe pain
Effect of VR-Distraction on pain | 15 minutes after 10 minute VR session.
  Pain scores will be collected. Pain will be rated using a numerical rating scale. Pain will be rated from 0 - 10. 0 meaning no pain 10 being severe pain
Effect of VR-Distraction on pain | 30 minutes after 10 minute VR session.
  Pain scores will be collected. Pain will be rated using a numerical rating scale. Pain will be rated from 0 - 10. 0 meaning no pain 10 being severe pain
Effect of VR-Biofeedback on anxiety | Before 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-Biofeedback on anxiety | Immediately after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-Biofeedback on anxiety | 15 minutes after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-Biofeedback on anxiety | 30 minutes after 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a numerical rating scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-Biofeedback on pain | Before 10 minute VR session
  Pain scores will be collected. Pain will be rated using a numerical rating scale. Pain will be rated from 0 - 10. 0 meaning no pain 10 being severe pain
Effect of VR-Biofeedback on pain | Immediately after 10 minute VR session
  Pain scores will be collected. Pain will be rated using a numerical rating scale. Pain will be rated from 0 - 10. 0 meaning no pain 10 being severe pain
Effect of VR-Biofeedback on pain | 15 minutes after 10 minute VR session
  Pain scores will be collected. Pain will be rated using a numerical rating scale. Pain will be rated from 0 - 10. 0 meaning no pain 10 being severe pain
Effect of VR-Biofeedback on pain | 30 minutes after 10 minute VR session
  Pain scores will be collected. Pain will be rated using a numerical rating scale. Pain will be rated from 0 - 10. 0 meaning no pain 10 being severe pain

SECONDARY OUTCOMES:
Role of anxiety on changes in pain | One time prior to study visit
  Participants will complete a questionnaire regarding anxiety
Role of pain catastrophizing | One time prior to study visit
  Participants will complete a questionnaire regarding pain

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Olbrecht, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
This information will be made available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available upon publication. All data will be deidentified.

REFERENCES:
- [Derived] Olbrecht VA, O'Conor KT, Williams SE, Boehmer CO, Marchant GW, Glynn SM, Geisler KJ, Ding L, Yang G, King CD. Guided Relaxation-Based Virtual Reality for Acute Postoperative Pain and Anxiety in a Pediatric Population: Pilot Observational Study. J Med Internet Res. 2021 Jul 12;23(7):e26328. doi: 10.2196/26328. PMID 34048358